CLINICAL TRIAL: NCT03127683
Title: The Influence of Head and Neck Position on Performance of Ambu AuraGainTM in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H1704-069-844
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2017-11

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Rotation

STUDY DESIGN:
Intervention Model Description: An AuraGain will be placed in all patients, and mechanical ventilation will be performed using a volume-controlled mode with a tidal volume of 10 ml/kg.
  The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed first for the neutral head position and then for the extended, flexed, and rotated head positions in a random order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AuraGain group (Experimental): An AuraGain will be placed in all patients, and mechanical ventilation will be performed using a volume-controlled mode with a tidal volume of 10 ml/kg.
  The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed first for the neutral head position and then for the extended, flexed, and rotated head positions in a random order.
  Interventions: Other: Neutral position; Other: Extension; Other: Flexion; Other: Rotation; Device: Ambu AuraGain TM

INTERVENTIONS:
Other: Neutral position — The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed at this position
  Other Names: Neutral position of head and neck
Other: Extension — The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed at this position
  Other Names: Head and neck extension
Other: Flexion — The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed at this position
  Other Names: Head and neck flexion
Other: Rotation — The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed at this position
  Other Names: Head and neck rotation
Device: Ambu AuraGain TM — Single Use Laryngeal Mask Sterile

SUMMARY:
The influence of different head and neck positions on the effectiveness of ventilation with the Ambu AuraGain airway remains unevaluated.

This study aimed to evaluate the influence of different head and neck positions on ventilation with the AuraGain airway.

An AuraGain will be placed in all patients, and mechanical ventilation will be performed using a volume-controlled mode with a tidal volume of 10 ml/kg.

The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed first for the neutral head position and then for the extended, flexed, and rotated head positions in a random order.

ELIGIBILITY:
Inclusion Criteria:

* Children < 7 years old who scheduled for general anesthesia using supraglottic airway

Exclusion Criteria:

* Children who require tracheal intubation
* Emergency operation without NPO
* History of C-spine surgery or disease
* History of Esophageal disease or surgery

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 30 seconds after positioning of head and neck
  The airway pressure at which a leak sound is detected around the patient's mouth and at which the airway pressure has reached equilibrium, when the pressure-limiting valve of the anesthesia breathing system is closed and the fresh gas flow rate was fixed at 3 L/min

SECONDARY OUTCOMES:
Peak inspiratory pressure | 30 seconds after positioning of head and neck
  peak airway pressure
Tidal volume | 30 seconds after positioning of head and neck
  Expiratory tidal volume
Fiberopic bronchoscopic view | 30 seconds after positioning of head and neck
  1. No visible glottis 2. Visible glottis and anterior epiglottis 3. Visible glottis and posterior epiglottis 4. Only visible glottis

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided